CLINICAL TRIAL: NCT01793909
Title: Role of Vascular Function: Oxygen Delivery vs Oxygen Utilization in the Exercise Impairment in Type 2 Diabetes
Brief Title: Type 2 Diabetes and Exercise Function in Single Leg Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-0062; 1564 (Other: Clinical Translational Research Center - University Hospital); 1UL1TR001082 (NIH)
Record Dates: First submitted 2012-12-11; First posted 2013-02-18 (Estimated); Results first posted 2019-05-20 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Exercise Impairment; Blood Flow; Muscle Oxygen Uptake; Exercise Training
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Leg Exercise (Other): Supervised single leg, exercise training of the index (dominant) calf muscle 5 days per week for two weeks - alternating weight-bearing single leg calf raises and single leg calf extensions by endurance resistance training (weight machine apparatus).
  Interventions: Other: Single Leg Exercise Training

INTERVENTIONS:
Other: Single Leg Exercise Training — Following the completion of baseline testing, all 3 subject groups will undergo supervised single leg, exercise training of the index (dominant) calf muscle 5 days per week for two weeks - alternating weight-bearing single leg calf raises and single leg calf extensions by endurance resistance training (weight machine apparatus).
  Other Names: Exercise Training

SUMMARY:
This study plans to learn more about the effects of type 2 diabetes (T2DM) on exercise blood flow and muscle oxygen uptake. This study will evaluate & compare exercise function during single leg plantar flexion exercise in a total of 45 subjects from the Denver area (15 lean controls, 15 people with T2DM, and 15 overweight control subjects).

Differences between the exercise responses in people with T2DM and healthy people will help further identify the disease process of T2DM and direct future research of treatments and interventions.

DETAILED DESCRIPTION:
It is well established that functional exercise capacity and peak oxygen uptake (VO2) are reduced in patients with type 2 diabetes mellitus (T2DM) compared with healthy counterparts. The mechanisms underlying the exercise deficit in T2DM remain largely unknown, but previous work has suggested that reduced exercise blood flow and impaired submaximal VO2 may be contributing factors. Both of these findings are consistent with a peripheral impairment of skeletal muscle oxygen delivery, oxygen utilization, or both. Indeed, dysfunction of skeletal muscle metabolism plays a key role in the pathophysiology of T2DM, and considerable work has described abnormalities of oxidative function in the skeletal muscle of people with T2DM. Given this, it is likely that the causes of exercise intolerance in T2DM may relate to specific defects at the level of the skeletal muscle, particularly given that skeletal muscle blood flow and oxidative capacity are impaired in diabetes. However, to our knowledge, no one has related these peripheral muscle abnormalities to the diminished exercise function in this patient group.

The overarching hypothesis for the proposed research is that both a failure to adequately increase muscle oxygen delivery following the onset of exercise and reduced oxidative function of skeletal muscle contribute to the acute oxygen deficit and diminished exercise tolerance that has been observed in patients with T2DM.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with and without type 2 diabetes
* 30-70 years of age
* Lean and overweight
* Sedentary subjects not participating in a regular exercise program (<one bout of exercise/week)

Exclusion Criteria:

* Documented cardiovascular disease
* Uncontrolled hypertension: systolic blood pressure (SBP) > 150, diastolic blood pressure (DBP)> 110
* Obstructive pulmonary disease or asthma
* Peripheral neuropathy
* Subjects taking beta blockers, insulin, or Thiazolidinediones (TZD)
* Current or past smoking within the last 2 years
* Anemia
* Control HbA1c > 6, T2DM HbA1c > 10
* Type 1 diabetes
* Any implanted metal in subject's body

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-06; Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judy Regensteiner, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Type 2 Diabetes: Individuals with a diagnosis of type 2 diabetes
- Overweight Controls: Individuals with a BMI 25-30 but otherwise healthy.
Period: Overall Study
Arm/Group | Type 2 Diabetes | Overweight Controls
Started | 30 | 25
Completed | 20 | 20
Not Completed | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Type 2 Diabetes | Overweight Controls | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 14 | 24
  >=65 years | 10 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (9) | 54 (12) | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 4 | 3 | 7
  White | 16 | 14 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 25 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Muscle Oxygen Saturation
Description: The investigators evaluated the dynamics of muscle deoxygenation (O2 extraction) using near infrared spectroscopy (NIRS) during single leg plantar flexion exercise to identify the predominant mechanisms of oxygen delivery versus oxygen utilization abnormalities in the muscle of T2DM during the transition from rest to exercise. These measurements were gathered continuously for 2-5 minutes of multiple exercise bouts within two visits, one prior to the exercise intervention period and one post exercise intervention.
Time Frame: 4.5 hrs each, pre- and post- Exercise Intervention
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Type 2 Diabetes | Overweight Controls
Number analyzed (Participants) | 14 | 13
percentage
  Pre-intervention | -10.7127 (6.07805) | -8.9149 (6.68906)
  Post-intervention | -12.471 (11.07039) | -8.7883 (7.49904)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the course of study participation, approximately 3-4 months for each participant. Overall adverse event data was collected through the entire study, lasting 8 years.
Arm/Group | Type 2 Diabetes | Overweight Controls
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 3/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Type 2 Diabetes (N=20) | Overweight Controls (N=20)
Elevated blood pressure during exercise (Vascular disorders) | 1 (1) | 0 (0)
Leg hematoma (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Leg hematoma secondary to muscle biopsy performed in study
Chest pain during exercise (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT01793909/Prot_SAP_000.pdf